CLINICAL TRIAL: NCT03984084
Title: The Biological Classification of Mental Disorders Study: Towards a New Taxonomy of Mental Disorders
Brief Title: Biological Classification of Mental Disorders
Acronym: BeCOME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Other Study IDs: 350-14
Record Dates: First submitted 2019-05-24; First posted 2019-06-12 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Mental Disorder; Depressive Disorder; Anxiety; Trauma and Stressor Related Disorders
Keywords: biomarkers; translational medical research; psychiatry; Research Domain Criteria (RDoC); omics; neuroimaging; taxonomy
MeSH Terms: conditions — Mental Disorders; Depressive Disorder; Anxiety Disorders; Trauma and Stressor Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood and saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- externally recruited participants: Self-referred affected and non-affected participants responding to advertisements
  Interventions: Other: no intervention
- In-house patients: Patients seeking treatment in the outpatient clinic of the Max-Planck-institute of Psychiatry
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
BeCOME intends to include at least 1000 individuals with a broad spectrum of affective, anxiety and stress-related mental disorders as well as 500 individuals unaffected by mental disorders. After a screening visit, all participants undergo in-depth phenotyping procedures and omics assessments on two consecutive days. Several validated paradigms (e.g., fear conditioning, reward anticipation, imaging stress test) are applied to stimulate a response in a basic system of human functioning (e.g., acute threat response, reward processing, stress response) that plays a key role in the development of affective, anxiety and stress-related mental disorders. The response to this stimulation is then read out across multiple levels. Assessments comprise omics, physiological, neuroimaging, neurocognitive, psychophysiological and psychometric measurements. The multilevel information collected in BeCOME will be used to identify data-driven biologically-informed categories of mental disorders using cluster analytical techniques. A subgroup of affected individuals (patients of the outpatients clinic of the Max Planck Institute of Psychiatry) are longitudinally observed regarding the stability of omics markers, vital parameters and symptom severity.

DETAILED DESCRIPTION:
Background:

A major research finding in the field of Biological Psychiatry is that symptom-based categories of mental disorders map poorly onto dysfunctions in brain circuits or neurobiological pathways. Many of the identified (neuro)biological dysfunctions are "transdiagnostic", meaning that they do not reflect diagnostic boundaries but are shared by different ICD/DSM diagnoses. The compromised biological validity of the current classification system for mental disorders impedes rather than supports the development of treatments that not only target symptoms but also the underlying pathophysiological mechanisms. The Biological Classification of Mental Disorders (BeCOME) study aims to identify biology-based classes of mental disorders that improve the translation of novel biomedical findings into tailored clinical applications.

Methods:

BeCOME intends to include at least 1000 affected individuals (recruited through advertisements/self-referral or visits in the institute's outpatient clinic or in collaborating practices) with a broad spectrum of affective, anxiety and stress-related mental disorders as well as 500 individuals unaffected by mental disorders (advertisements/self-referral). After a screening visit, all participants undergo in-depth phenotyping procedures and omics assessments on two consecutive days. Several validated paradigms (e.g., fear conditioning, reward anticipation, imaging stress test) are applied to stimulate a response in a basic system of human functioning (e.g., acute threat response, reward processing, stress response) that plays a key role in the development of affective, anxiety and stress-related mental disorders. The response to this stimulation is then read out across multiple levels. Assessments comprise omics, physiological, neuroimaging, neurocognitive, psychophysiological and psychometric measurements. The multilevel information collected in BeCOME will be used to identify data-driven biologically-informed categories of mental disorders using cluster analytical techniques. Moreover, the subgroup of patients from the outpatient clinic of the Max Planck Institute of Psychiatry is followed-up at study days 14, 28 and 56 as well as 4 and 12 months after baseline for changes in a subset of parameters (omics, vital parameters and selected psychometric measures).

Discussion:

The novelty of BeCOME lies in the dynamic in-depth phenotyping and omics characterization of individuals with mental disorders from the depression and anxiety spectrum of varying severity. The investigators believe that such biology-based subclasses of mental disorders will serve as better treatment targets than purely symptom-based disease entities, and help in tailoring the right treatment to the individual patient suffering from a mental disorder. BeCOME has the potential to contribute to a novel taxonomy of mental disorders that integrates the underlying pathomechanisms into diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an affective, anxiety or stress-related mental disorder according to the criteria of DSM-IV or DSM-5 (Depressive disorders;Anxiety and obsessive-compulsive disorders: agoraphobia with and without panic disorder, panic disorder, social phobia, specific phobia, generalized anxiety disorder, obsessive compulsive disorder; Stress and trauma-associated mental disorders (e.g. posttraumatic stress disorder).
* or no mental disorder

Exclusion Criteria:

* Intake of any psychotropic medication/substance for a minimum of 2 months before study day 1.
* Current illness in the field of organic mental disorders;
* Affective disorders caused by a medical condition
* Organic mental disorders (e.g. dementia)
* Current disorders of schizophrenia;
* Current eating disorder;
* Mental retardation and profound developmental disorders;
* Severe neurological or internal medical illness;
* Posttraumatic or post-ischemic brain damage or elapsed cerebral hemorrhage;
* Acute suicidality;
* Pregnancy and postpartum period;
* Magnetic resonance imaging contraindications (e.g. non-MR compatible metal implants including cardiac pacemakers, claustrophobia);
* Myopia <-6 D, which cannot be compensated by contact lenses or MR compatible glasses (Cambridge Research Systems, Rochester, UK);
* Current substance abuse;
* Current or past substance dependence;
* Risky alcohol consumption, screened with the Alcohol Use Disorder Identification Test - Consumption questions (AUDIT-C) and defined as score of ≥5 in males and of ≥4 in females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with varying degrees and a broad range of mental disorders from the anxiety and depression spectrum
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-06-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of data-driven biologically-informed categories ("biotypes") of anxiety, depressive and stress-related mental disorders | cross-sectional (baseline)
  The study is exploratory. Following an Research Domain Criteria (RDoC) approach, the study will use multi-level information for clustering of patients anxiety, depressive and stress-related mental disorders.
Comparison of the new biotypes (biological classification approach) to traditional symptom-based diagnostic categories (DIA-X/M-CIDI) | cross-sectional (baseline)
  Assessment of anxiety, depressive and stress-related disorders using the diagnostic interview (computerized Munich version of the Composite International Diagnostic Interview, DIA-X/M-CIDI) according to the traditional classification approach in order to assess the distribution of "biotypes" across traditional diagnostic categories of affective and anxiety disorders.

OTHER OUTCOMES:
Stability/change in methylation over time | baseline and at days 14, 28 and 56 after baseline
  longitudinal analysis only in patients who are treated at the MPIP (group 2), DNA extraction from blood for the determination of epigenetic markers (DNA methylation) for the determination of the stability of methylation patterns from baseline up to study day 56.
Stability/change in body mass index (BMI) over time | baseline and at day 56 after baseline
  longitudinal analysis only in patients who are treated at the MPIP (group 2), comparison of body mass index (BMI, calculated as kg/m^2) at study day 56 to body mass index at baseline
Stability/change in blood pressure over time | baseline and at days 14, 28 and 56 after baseline
  longitudinal analysis only in patients who are treated at the MPIP (group 2), changes of blood pressure between baseline and study day 56.
Stability/change in gene expression over time | baseline and at days 14, 28 and 56 after baseline
  longitudinal analysis only in patients who are treated at the MPIP (group 2), messenger RNA extraction from blood for the determination of changes in gene expression from study day 1 up to study day 56.
Stability/change in BDI-II (Beck-Depression-Inventory-II) sum score | baseline and every follow-up assessment: day 14, 28 and 56 as well as 4 and 12 months after baseline)
  longitudinal analysis only in patients who are treated at the MPIP (group 2), Beck depression inventory, revised version (BDI-II) will be used for the assessment of changes in depression severity (indicated by the sum score, range from 0 to 63) from study day 1 up to 12 months after study day 1
Stability/change in the Montgomery Asberg Depression Scale (MADRS) sum score | baseline and every follow-up assessment: day 14, 28 and 56 as well as 4 and 12 months after baseline)
  longitudinal analysis only in patients who are treated at the MPIP (group 2), the observer-based Montgomery Asberg Depression Scale (MADRS) will be used for the assessment of changes in MADRS depression sum score (range from 0 to 60) from study day 1 up to 12 months after study day 1
Stability/change in the state scale of the Spielberger State-Trait Anxiety Inventory (STAI) | baseline and every follow-up assessment: day 14, 28 and 56 as well as 4 and 12 months after baseline)
  longitudinal analysis only in patients who are treated at the MPIP (group 2), the sum score of the state scale of the STAI (range from 20 to 80) will be used for the assessment of changes in state anxiety from study day 1 up to 12 months after study day 1
Stability/change in the Panic and Agoraphobia Scale (PAS) score over time | baseline and every follow-up assessment: day 14, 28 and 56 as well as 4 and 12 months after baseline)
  longitudinal analysis only in patients who are treated at the MPIP (group 2), the sum score of Panic and Agoraphobia Scale (PAS), range from 0 to 65, will be used for the assessment of changes in the severity of panic and agoraphobia.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Binder, Prof. Dr. Dr., Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun R, Fietz J, Erhart M, Poehlchen D, Henco L, Bruckl TM; BeCOME study team; Czisch M, Saemann PG, Spoormaker VI. Free-viewing gaze patterns reveal a mood-congruency bias in MDD during an affective fMRI/eye-tracking task. Eur Arch Psychiatry Clin Neurosci. 2024 Apr;274(3):559-571. doi: 10.1007/s00406-023-01608-8. Epub 2023 Apr 23. PMID 37087709
- [Derived] Bruckl TM, Spoormaker VI, Samann PG, Brem AK, Henco L, Czamara D, Elbau I, Grandi NC, Jollans L, Kuhnel A, Leuchs L, Pohlchen D, Schneider M, Tontsch A, Keck ME, Schilbach L, Czisch M, Lucae S, Erhardt A, Binder EB. The biological classification of mental disorders (BeCOME) study: a protocol for an observational deep-phenotyping study for the identification of biological subtypes. BMC Psychiatry. 2020 May 11;20(1):213. doi: 10.1186/s12888-020-02541-z. PMID 32393358